CLINICAL TRIAL: NCT01059214
Title: Cardiac MRI for Patients Enrolled in INFUSE-AMI
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100034; 10-H-0034
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2012-10-11

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease; Myocardial Fibrosis; Gadolinium; Myocardial Edema
Keywords: Acute Myocardial Infarction; Reperfusion; MRI; Heart Attack
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* INFUSE AMI is an ongoing clinical trial examining how patients with heart attacks are treated. The study's aim is to help determine the best way to treat patients with specific kinds of heart attacks caused by blood clots.
* To evaluate the effect of the heart attack on the heart tissue and function, participants in the INFUSE-AMI study will have magnetic resonance imaging (MRI) scans of the heart at specific times after their heart attack.

Objectives:

- To perform cardiac MRI scans on patients who are participating in the INFUSE-AMI study.

Eligibility:

- Individuals at least 18 years of age who are enrolled in the INFUSE-AMI study.

Design:

* Participants will have an MRI scan of the heart about 5 days and between 23 and 44 days after their heart attack. The MRI scan at day 5 is optional.
* Participants will provide a blood sample prior to the MRI scan.
* During the scan, participants will be given a contrast drug to show the blood flow to and within the heart. An electrocardiogram will be used to monitor the heart during the procedure.
* No other treatment will be provided in this protocol.

DETAILED DESCRIPTION:
The purpose of this research protocol is to perform contrast enhanced cardiac MRI studies on patients enrolled in the INFUSE-AMI study (INFUSE-AMI is a multicenter, open-label controlled single-blind randomized study with up to 452 patients enrolled in approximately 50 US and European sites). Patients who present with anterior ST elevation myocardial infarction by electrocardiogram (STEMI) and an occluded proximal or mid left anterior descending artery (LAD) with TIMI 0/1 flow will be eligible for randomization to one of the following arms: 1) Local infusion of Abciximab and thrombus aspiration, 2) Local infusion of Abciximab and no thrombus aspiration, 3) No local infusion and thrombus aspiration, or 4) No local infusion and no thrombus aspiration. Cardiac MRI is performed to assess left ventricular function and infarct size for the primary INFUSE-AMI study. Thus, this local research protocol will provide the cardiac MRI scans at no cost to the participant. Additional images of the heart will be obtained for local research purposes. Cardiac MRI scans will be performed at around 5 days (optional) and at 30 days after myocardial infarction.

ELIGIBILITY:
-INCLUSION CRITERIA:

i. Signed consent for INFUSE-AMI

ii. Ability to travel to the NIH for participation in MRI studies. and

iii. Ability to provide informed consent, or holds a valid surrogate decision maker authorization (such as Durable Power of Attorney).

EXCLUSION CRITERIA:

i. Known hypersensitivity or contraindication to gadolinium contrast

ii. Severe kidney disease (eGFR <30 mLIminIl .73 m(2) BSA)

iii. Pregnancy

iv. Breast feeding (unless subject is willing to discard breast milk for 24 hours)

v. Cardiac pacemaker or implantable defibrillator

vi. Non-MRI compatible aneurysm clip

vii. Neural stimulator (e.g. TENS unit)

viii. Any implanted or magnetically activated device (e.g. insulin pump)

ix. Any type of non-MRI compatible metallic ear implant

x. Metal shavings in the orbits

xi. Any metallic or foreign body, shrapnel, or bullet in a location which the physician feels would present a risk to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2009-12-10; Study Completion 2012-10-11

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Arai, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Frank JA, Mattay VS, Duyn J, Sobering G, Barrios FA, Zigun J, Sexton R, Kwok P, Woo J, Moonen C, et al. Measurement of relative cerebral blood volume changes with visual stimulation by 'double-dose' gadopentetate-dimeglumine-enhanced dynamic magnetic resonance imaging. Invest Radiol. 1994 Jun;29 Suppl 2:S157-60. doi: 10.1097/00004424-199406001-00052. No abstract available. PMID 7928216
- [Background] Mattay VS, Weinberger DR, Barrios FA, Sobering GS, Kotrla KJ, van Gelderen P, Duyn JH, Sexton RH, Moonen CT, Frank JA. Brain mapping with functional MR imaging: comparison of gradient-echo--based exogenous and endogenous contrast techniques. Radiology. 1995 Mar;194(3):687-91. doi: 10.1148/radiology.194.3.7862963.
- [Background] Deo A, Fogel M, Cowper SE. Nephrogenic systemic fibrosis: a population study examining the relationship of disease development to gadolinium exposure. Clin J Am Soc Nephrol. 2007 Mar;2(2):264-7. doi: 10.2215/CJN.03921106. Epub 2007 Feb 7. PMID 17699423